CLINICAL TRIAL: NCT02090725
Title: Controlled Trial of 3,4-Diaminopyridine in LEMS
Brief Title: Controlled Trial of 3,4-Diaminopyridine (3-4DAP) in Lambert-Eaton Myasthenic Syndrome (LEMS)
Acronym: 3-4DAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug receive FDA approval
Sponsor: Jeffrey A. Cohen, MD (Other)
Collaborators: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey A. Cohen, MD, Neurology Department Chair, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D04013
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Muscle Weakness
Keywords: fluctuating muscle weakness; hyporeflexia; autonomic Dysfunction
MeSH Terms: conditions — Muscle Weakness; Reflex, Abnormal; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3-4 Diaminopyridine (DAP) (Experimental)
  Interventions: Drug: 3-4 Diaminopyridine

INTERVENTIONS:
Drug: 3-4 Diaminopyridine
  Other Names: 3-4 DAP

SUMMARY:
The main purpose for this study is to provide access to 3,4 DAP, a drug which has demonstrated to be effective in treating weakness associated with Lambert-Eaton Myasthenic Syndrome. LEMS is a rare autoimmune cause of a defect in neuromuscular transmission. The disorder is clinically characterized by fluctuating muscle weakness, hyporeflexia and autonomic dysfunction.

DETAILED DESCRIPTION:
More than half of LEMS cases are associated with malignancy, usually small cell lung cancer. These paraneoplastic cases progress more quickly than primary autoimmune LEMS. An overlap syndrome with other autoimmune diseases is often detected in LEMS patients.

3,4 DAP is effective in LEMS because it increases calcium influx into the nerve terminal by blocking potassium efflux and thereby prolonging the presynaptic action potential. 3,4 DAP is less likely to provoke epileptic seizures than its precursor, 4-aminopyridine, because it is less able to cross the blood-brain barrier. 3,4 DAP is effective in increasing strength and improving autonomic symptoms in LEMS patients of both the primary autoimmune and paraneoplastic etiologies.

ELIGIBILITY:
Inclusion Criteria: -Male or female majority between 45 and 60 years of age

* diagnosed with Lambert-Eaton Myasthenic Syndrome.
* subjects must be taking full dose of pyridostigmine

Exclusion Criteria: - does subject have a history of liver problems?

* does subject have a history of prolonged QTc syndrome (which is a condition where there is prolongation between the start of the Q wave and the end of the T wave in the heart's electrical cycle).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-02; Primary Completion 2018-07 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Cohen, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3-4 Diaminopyridine (DAP): 3-4 Diaminopyridine
  Treatment will begin with 5mg three time a day. A common final dosage is 15mg four or five time a day, as clinically needed, and if tolerated. The upper limit is a total of 100mg/day.
Period: Overall Study
Arm/Group | 3-4 Diaminopyridine (DAP)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — participants moved from area | 3

BASELINE CHARACTERISTICS:
Groups:
- 3-4 Diaminopyridine (DAP): 3-4 Diaminopyridine
Arm/Group | 3-4 Diaminopyridine (DAP)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Showed Improvement in Muscle Weakness During Their Last Study Related Visit
Description: Muscle weakness will be assessed monthly for the first 3 months based on clinical assessment during office visits. Muscle weakness will then be assessed every 6 months once the patient is stabilized based on clinical assessments during office visits. The assessment of whether there was an improvement in muscle weakness, based on the PI's clinical judgment, was noted during the last study visit completed by the participant.
Time Frame: Participants were followed until they withdrew or the study ended. Time frame ranged from 1 month to 3 years.
Population: One participant was not on the study long enough to complete the one month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 3-4 Diaminopyridine (DAP)
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Participants were followed until they withdrew from the trial. Adverse events were evaluated at Month 1, Month 2, Month 3, then every 6 months once patient is stable. The total time period over which adverse events were evaluated ranged from 2 weeks to 3 years.
Arm/Group | 3-4 Diaminopyridine (DAP)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2008-09-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT02090725/Prot_000.pdf